CLINICAL TRIAL: NCT01050842
Title: Pilot Trial to Evaluate the Safety and Efficacy of the Administration of Bicalutamide (Casodex TM) Per Day in Combination With Raloxifene (Evista TM) Per Day in Patients With Hormone Refractory Prostate Cancer
Brief Title: Bicalutamide and Raloxifene in Treating Patients With Metastatic or Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0851; NCI-2009-01700 (Registry Identifier: NCI-CTRP); 07-008912 (Other: Mayo IRB); MC0851 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2016-03

CONDITIONS: Prostate Cancer; Adenocarcinoma of the Prostate; Hormone-resistant Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Raloxifene Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral bicalutamide and oral raloxifene on days 1-28.
  Interventions: Drug: bicalutamide; Drug: raloxifene; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: bicalutamide — Given orally
  Other Names: Casodex; CDX; Cosudex; ICI 176,334
Drug: raloxifene — Given orally
  Other Names: Evista; Keoxifene; LY 139481; RALOX
Procedure: quality-of-life assessment — Ancillary study
  Other Names: quality of life assessment

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as bicalutamide, may lessen the amount of androgens made by the body. Selective estrogen receptor modulators, such as raloxifene, may work together with bicalutamide to stop the growth of prostate cancer.

PURPOSE: This clinical trial studies giving bicalutamide and raloxifene together in treating patients with metastatic or hormone-refractory prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To describe the 6-month progression-free survival rate, progression-free survival, and overall survival of patients receiving bicalutamide and raloxifene.

II. To describe the adverse event profile of combined treatment with bicalutamide and raloxifene (adverse events graded using the NCI CTCAE version 3.0).

III. To describe the quality of life of patients receiving bicalutamide and raloxifene.

OUTLINE: Patients receive oral bicalutamide and oral raloxifene on days 1-28. Treatment repeats for up to 6 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed every 3-6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of prostate adenocarcinoma
* Objective disease progression or rising PSA despite androgen deprivation therapy
* Progression of measurable disease assessed within 28 days prior to registration; progression of non-measurable disease assessed within 28 days prior to registration; patients with rising PSA must demonstrate a rising trend with two successive elevations at a minimum interval of two weeks
* Patients must have been surgically or medically castrated; if the method of castration is LHRH agonists (leuprolide or goserelin) or LHRH antagonists, then the patient should be willing to continue the use of LHRH agonists; castration using LHRH agonist should not be interrupted and patients who have stopped treatment should be willing to restart
* If the patient has been treated with non-steroidal antiandrogens (bicalutamide, flutamide, nilutamide, or ketoconazole) then they must have stopped at least 14 days prior to registration for ketoconazole and at least 28 days prior to registration for bicalutamide, flutamide, or nilutamide and the patients must have demonstrated progression
* Any patient with documented antiandrogen withdrawal syndrome with bicalutamide would not be eligible
* A minimum PSA of 5 ng/ml or new areas of bony metastases on bone scan are required for patients with no measurable disease; no minimum PSA requirement for patients with measureable disease
* ECOG Performance Status (PS) 0, 1, or 2
* ANC >= 1500
* PLT >= 100,000
* HgB >= 9.0 g/dL
* Total bilirubin =< 1.5 x UNL
* SGOT (AST) =< 3 x UNL
* SGPT (ALT) =< 3 x UNL
* Alkaline Phosphatase =< 3 x UNL
* Creatinine =< 1.5 x UNL
* Ability to complete questionnaire(s) independently or with assistance
* Provide informed written consent
* Willingness to return to Mayo Clinic enrolling institution for follow-up

Exclusion Criteria:

* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients with known HIV infection
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Prior radiation therapy is allowed; at least 21 days must have elapsed since completion of radiation therapy, and patients must have recovered from side effects
* Patients may have received prior surgery; at least 21 days must have elapsed since completion of surgery and patient must have recovered from all side effects
* The use of bisphosphonates is allowed provided that the patient has been receiving that medication for >= 4 weeks with evidence of progressive disease
* Prior systemic therapy to treat prostate cancer including cytotoxic chemotherapy, biologic therapy, vaccine therapy, and experimental therapy is allowed, and at least 28 days must have elapsed since completion of therapy and the patient must have recovered from all side effects
* No concurrent use of estrogen, estrogen-like agents, or other hormonal therapy is allowed; prior use of these agents will need to be discontinued >= 4 weeks prior to registration
* Active other malignancy, except non-melanotic skin cancer or carcinoma-in-situ of the cervix; if there is a history of prior malignancy, must not be receiving other specific treatment (other than hormonal therapy) for cancer
* History of congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Experienced documented anti-androgen withdrawal syndrome on bicalutamide
* History of venous thromboembolic disease or significant risk for venous thromboembolic disease
* History of symptomatic coronary artery disease
* History of stroke or significant risk for stroke

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2012-10-04 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate | 6 months
Adverse events of combined treatment with bicalutamide and raloxifene as measured by CTCAE version 3.0
Quality of life as assessed by Linear Analogue Self Assessment (LASA6) and the Hormonal Domain scale of the Expanded Prostate Cancer Index Composite (EPIC-H) survey
Survival time
Measurable or evaluable disease as assessed by RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Erik P. Castle, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic In Arizona, Scottsdale, Arizona, United States